CLINICAL TRIAL: NCT02296463
Title: A Phase I Randomized, Observer-Blinded, Dose-Ranging Study to Evaluate the Immunogenicity and Safety of a Respiratory Syncytial Virus (RSV) Recombinant Fusion (F) Nanoparticle Vaccine, With or Without Aluminum Adjuvant, in Healthy Subjects 24 to <72 Months of Age
Brief Title: A Phase I Randomized, Observer-Blinded, Dose-Ranging Study in Healthy Subjects 24 to <72 Months of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RSV-P-101
Record Dates: First submitted 2014-11-08; First posted 2014-11-20 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Respiratory Synctial Virus
MeSH Terms: interventions — Adjuvants, Pharmaceutic; Injections; Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment Group A (Experimental): Day 0: RSV F Vaccine with adjuvant, Day 28: RSV F Vaccine with adjuvant
  Interventions: Biological: RSV F Vaccine with adjuvant (0.5mL injection)
- Treatment Group B (Experimental): Day 0: RSV F Vaccine with adjuvant, Day 28: Hepatitis A Vaccine
  Interventions: Biological: RSV F Vaccine with adjuvant (0.5mL injection); Biological: Hepatitis A Vaccine (0.5mL injection)
- Treatment Group C (Experimental): Day 0: RSV F Vaccine, Day 28: RSV F Vaccine
  Interventions: Biological: RSV F Vaccine (0.5mL injection)
- Treatment Group D (Experimental): Day 0: RSV F Vaccine, Day 28: Hepatitis A Vaccine
  Interventions: Biological: RSV F Vaccine (0.5mL injection); Biological: Hepatitis A Vaccine (0.5mL injection)
- Treatment Group E (Placebo Comparator): Day 0: Placebo, Day 28: Hepatitis A Vaccine
  Interventions: Biological: Hepatitis A Vaccine (0.5mL injection); Biological: Placebo (0.5mL injection)

INTERVENTIONS:
Biological: RSV F Vaccine with adjuvant (0.5mL injection)
  Arms: Treatment Group A; Treatment Group B
Biological: RSV F Vaccine (0.5mL injection)
  Arms: Treatment Group C; Treatment Group D
Biological: Hepatitis A Vaccine (0.5mL injection)
  Arms: Treatment Group B; Treatment Group D; Treatment Group E
Biological: Placebo (0.5mL injection)
  Arms: Treatment Group E

SUMMARY:
This is a randomized, observer-blind, irrelevant comparator-controlled trial in male and female subjects ≥24 months of age and <72 months of age. Subjects will be without symptomatic chronic cardiopulmonary disease, including recurrent wheezing. Subjects will be screened for seropositivity to RSV in a qualified serum microneutralization (MN) assay and will be excluded if titers for either RSV/A or RSV/B are <1:16 (4 log2).

Treatments will comprise an IM dose of saline placebo or RSV F vaccine on Day 0 and an IM dose of RSV F vaccine or a licensed hepatitis A vaccine on Day 28. Hepatitis A vaccine (and in one group placebo) will be used to maintain the study blind; all subjects will receive a complete course of hepatitis A vaccine as a study benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females, ≥24 months of age and <72 months of age, without known chronic cardiopulmonary disease including especially persistent or frequently recurrent wheezing.
2. Free of other illnesses that are believed to increase the risks associated with influenza or other respiratory viral infections, including: diabetes mellitus, congenital or acquired blood dyscrasias, renal or hepatic dysfunction, and morbid obesity.
3. Parent(s)/guardian(s) willing and able to give informed consent prior to study enrollment, and assert ability to comply with study requirements.
4. Parent(s)/guardian(s) and/or other designated child care provider must have continuous capacity for telephone communication with the study site.

Exclusion Criteria:

1. Serum MN titers against RSV/A or RSV/B <1:16 (4 log2).
2. Toxicity grade ≥2 for any safety laboratory parameter.
3. Participation in research involving an investigational product (drug/biologic/device) within 45 days before planned date of first vaccination and planned participation at any time during the study.
4. History of a serious reaction to any prior vaccination, including Guillain-Barré Syndrome within six weeks following a previous influenza vaccination.
5. Receipt of any vaccine (other than the influenza vaccine specified in the protocol) in the four weeks preceding the first study vaccination and/or planned receipt of a licensed vaccine (other than the hepatitis A vaccine specified in the protocol) at any time prior to Study Day 56.
6. Receipt of an RSV vaccine at any time.
7. Any known or suspected immunosuppressive condition, acquired or congenital, as determined by medical history and/or physical examination.
8. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccine. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose ≥1 mg/kg of prednisone per day or equivalent. The use of topical glucocorticoids for minor cutaneous symptoms will be permitted, but the use of nasal or inhaled glucocorticoids in exclusionary (because of potential related diagnoses rather than immunosuppression).
9. Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or during the study.
10. Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever or an oral temperature >38.0°C on the planned day of vaccine administration).
11. Known disturbance of coagulation.
12. Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled or could interfere with evaluation of the vaccine or interpretation of study results (including social, neurologic, or psychiatric conditions in the subject or parent(s)/guardian(s) deemed likely to impair the quality of safety reporting).

Ages: 24 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2014-11; Primary Completion 2015-09 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Numbers and percentages of subjects with solicited local and systemic AEs. | Up to Day 392
  Solicited local and systemic AEs over the 7 days post injection; and all AES, solicited and unsolicited, including adverse changes in clinical laboratory parameters, over 56 days post- first injection. In addition, MAEs, SAEs, and SNMCs will be collected for one year.
Immunogenicity as assessed by serum IgG antibody levels specific for the F protein antigen as detected by enzyme-linked immunosorbent assay (ELISA) providing a standardized ELISA Unit (EU) reasout based on a standard reference sample. | Up to Day 392
  Derived/ calculated endpoints based on these data will include:
  Geometric mean EU (GMEU) Geometric mean ratio (GMR) Seroresponse rate (SRR)

SECONDARY OUTCOMES:
Epitope-specific immune responses to the RSV F protein antigen measured by serum titers in a competition ELISA assay using known-efficacious prophylactic antibody preparation, or in vitro neutralization assays using at least one prototype RSV/A and RSV/B | Up to Day 392
  Derived/ calculated endpoints based on these data will include:
  Geometric mean EU (GMEU) Geometric mean ratio (GMR) Seroconversion rate (SCR) Seroresponse rate (SRR)

OTHER OUTCOMES:
Epitope-specific immune responses to the RSV F protein antigen measured by serum titers in a direct binding ELISA using an immobilized linear peptide representing the conserved RSV F protein neutralizing antigenic site II. | Up to Day 392
  Derived/ calculated endpoints based on these data will include:
  Geometric mean EU (GMEU) Geometric mean ratio (GMR) Seroconversion rate (SCR) Seroresponse rate (SRR)

CONTACTS AND LOCATIONS:
Overall Officials: D. Nigel Thomas, Ph.D., Study Director — Novavax
Locations (4):
- Canada (4):
  - University of Calgary, Alberta Children's Hospital, Calgary, Alberta
  - Dalhousie University, IWK Health Centre- Canadian Center for Vaccinology, Halifax, Nova Scotia
  - Aggarwal and Associates, Brampton, Ontario
  - Medicore Research, Inc, Greater Sudbury, Ontario

REFERENCES:
- See also: Related Info — http://www.novavax.com